CLINICAL TRIAL: NCT02143674
Title: MUSCLE STRENGTHENING EXERCISES AND GLOBAL STRETCHING: IMPACT ON BALANCE, FEAR OF FALLING AND FUNCTIONAL CAPACITY OF ELDERLY
Brief Title: Muscle Strengthening Exercises and Global Stretching in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria das Graças Rodrigues de Araújo, PhD, Universidade Federal de Pernambuco
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFPernambuco; UFPE CAAE N.130.281 (Other: UFPE CAAE N.130.281)
Record Dates: First submitted 2014-02-27; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Osteoporosis; Senile Osteopenia
Keywords: Stretching exercise muscle; Elderly; Techniques and exercise; Physiotherapy
MeSH Terms: conditions — Osteoporosis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INTERVENTION (Experimental): Muscle stretching and Strength Training
  Interventions: Other: Muscle stretching and Strength Training
- Educated about physical exercises (Experimental)
  Interventions: Other: Educated about physical exercises

INTERVENTIONS:
Other: Muscle stretching and Strength Training — Each step of stretching on specific muscles was repeated three times by keeping the posture for 30 seconds, (Arnold and Kokkonen, 2007; Toraman A, Yildirim. 2010; Dai, Ware, Giuliani, 2012; Duque et al., 2013; Granacher et al., 2013). The Pectoral, Quadriceps, Paraspinal, Abdominal and Ischial tibial and sural triceps muscles were elongated.
  Strength Training Muscle strengthening was performed using weights and dumbbells. The training load individually determined through the test of strength with 10 repetitions maximum. The load was reevaluated four weeks of training. The Abdominal, Paraspinal, Quadriceps and Posterior thigh muscles (hamstrings) were submitted to the intervention protocol.
  Arms: INTERVENTION
Other: Educated about physical exercises
  Arms: Educated about physical exercises

SUMMARY:
Introduction: The life expectancy and the number of people hitting the old age have increased in recent years. The aging process is accompanied by morphological and functional changes that contribute to reduced functional capacity, increase the number of falls and the appearance of physical limitations. Exercise promotes maintenance of functional autonomy, improving the physical ability of the elderly making it more independent.

Objective: To evaluate the effect of a program of muscle strengthening exercises associated with global stretching on balance, fear of falling and functional capacity in elderly women.

Methods: This was a non-randomized controlled trial, in which 12 volunteers aged over 60 years were divided into two groups: intervention group (IG, n = 7) submitted to muscle strengthening exercises and stretching, 2 times per week for 12 weeks, and the control group (CG, n = 5), not submitted to the protocol but were educated about physical exercises. Before and after the protocol were evaluated scores of Berg Balance Scale, the Falls Efficacy Scale International (FES-I) and Evaluation of Functional Autonomy Development Group for Latin American Maturity (GDLAM). Data were statistically analyzed within and between groups with a significance level of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* women aged over 60 years,
* independent in locomotion,
* with ability to understand verbal commands to perform the tests and participation in the treatment program

Exclusion Criteria:

* execution of other physical activities or doing other types of physical therapy,
* had any prior neurological deficit (stroke, traumatic brain injury, Parkinson's disease) or
* musculoskeletal diseases which compromising performance and mobility,
* use of orthosis for locomotion,
* inability to perform the evaluation tests and/or participation in the intervention session

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
balance score | 12 weeks
  Berg Balance Scale (BBS)

SECONDARY OUTCOMES:
Fear of falling score | 12 weeks
  Falls Efficacy Scale International (FES-I)
Functional Capacity | 12 weeks
  Evaluation of the Latin American Functional Autonomy Development Group for Maturity (GDLAM)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Kinesiotherapy and Manual Therapeutic Resources, Department of Physical Therapy, Federal University of Pernambuco (UFPE), Recife, Pernambuco, Brazil